CLINICAL TRIAL: NCT07064148
Title: The Effects of Self-Myofascial Release on Physical Fitness and Swing Performance in Male Collegiate Golfers in China
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Qi (Other)
Responsible Party: Sponsor-Investigator, Yang Qi, Doctoral Researcher, Department of Sports Studies, Universiti Putra Malaysia, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025011
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Range of Motion, Articular; Physical Fitness; Golf Specific Performance
Keywords: Golf; Physical fitness; swing performance

STUDY DESIGN:
Intervention Model Description: This study employed a parallel-group randomized controlled trial design with two arms: an intervention group receiving self-myofascial release (SMR) and a passive control group. Participants were randomly assigned in a 1:1 ratio using a computer-generated sequence. All participants underwent a centralized 3-month training program with identical routines, meals, and accommodations. The intervention lasted 8 weeks. The SMR group received supervised sessions three times per week (30 minutes/session) in the evening after regular training. The control group engaged in time-matched passive video viewing to control for attention bias. Randomization and timing were standardized, and outcome assessors were blinded to group allocation.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation throughout the study. All participants were assigned ID codes, and test results were recorded without any indication of group assignment. Assessors were not involved in the delivery of the intervention or in regular training sessions, and all assessments (physical fitness and swing performance) were conducted in a standardized manner to reduce potential bias. The blinding process was maintained until data analysis was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Myofascial Release (SMR) Group (Experimental): The SMR program was delivered three times per week (Mondays, Wednesdays, and Fridays), each session lasting approximately 30 minutes and conducted after 7:00 PM in the on-site gym, immediately following daily golf training. Prior to the first session, a certified instructor provided standardized instruction on SMR techniques using foam rollers and massage balls targeting the thoracolumbar fascia, gluteal and hip complex, hamstrings, and shoulder girdle. All sessions were supervised to ensure compliance and correct execution. SMR exercises were performed in a fixed sequence. All participants in the SMR group used the same model of equipment purchased in bulk from Decathlon (DOMYOS brand), including a 45 cm × 15 cm high-density EVA foam roller and a 6.5 cm massage ball. Participants in the SMR group did not engage in any video watching activities during the intervention period, unlike the control group.
  Interventions: Behavioral: Self-Myofascial Release (SMR) Program
- Control Group (No SMR) (Sham Comparator): Participants in the control group did not receive any self-myofascial release (SMR) intervention. They followed the same daily training schedule, accommodation, and meals as the SMR group. Instead of SMR, they engaged in supervised viewing of golf-related instructional videos or documentaries three times per week, approximately 30 minutes per session, after 7:00 PM in a designated classroom. This was matched in timing and frequency to the SMR group's sessions. No flexibility, mobility, or soft tissue techniques were included. Sessions were conducted collectively at the same time and setting as the SMR group to control for attention and environmental bias. Attendance and compliance were monitored by supervisors.
  Interventions: Behavioral: Golf-Related Video Viewing (Attention Control)

INTERVENTIONS:
Behavioral: Self-Myofascial Release (SMR) Program — The intervention involves a structured 6-week Self-Myofascial Release (SMR) program using foam rollers and massage balls. Participants perform standardized SMR exercises targeting major muscle groups relevant to golf performance, including the calves, hamstrings, glutes, back, shoulders, and thoracic spine. The intervention is conducted three times per week, with each session lasting approximately 30 minutes. Exercises are demonstrated and monitored by certified instructors. The control group continues regular physical activities without SMR.
  Arms: Self-Myofascial Release (SMR) Group
Behavioral: Golf-Related Video Viewing (Attention Control) — Participants in the control group did not receive any self-myofascial release (SMR) intervention. They followed the same daily training schedule, accommodation, and meals as the SMR group. Instead of engaging in SMR exercises, participants in the control group engaged in supervised viewing of golf-related instructional videos or documentaries three times per week, approximately 30 minutes per session, after 7:00 PM in a designated classroom. This viewing schedule was matched in timing and frequency to the SMR group's intervention sessions. No flexibility, mobility, or soft tissue techniques were included in the control group's activities. The sessions were conducted collectively in the same setting and at the same time as the SMR group to control for attention and environmental bias. Attendance and compliance were closely monitored by supervisors to ensure adherence.
  Arms: Control Group (No SMR)

SUMMARY:
This is a randomized controlled trial aimed at evaluating the effects of a self-myofascial release (SMR) program on physical fitness and swing performance in male collegiate golfers in China. The primary purpose is to determine whether SMR, using foam rollers and massage balls, can improve joint mobility, core control, balance, and golf-specific swing outcomes.

The study seeks to answer the following key questions:

Can an 8-week SMR program enhance physical functions such as mobility, balance, and trunk control in male collegiate golfers?

Can SMR improve key performance indicators of golf swing, including club head speed, ball speed, carry distance, and accuracy?

Participants (n=60) will be healthy male collegiate golfers aged 18-25, randomly assigned to either an experimental group (SMR) or a time-matched control group (no SMR). Both groups will undergo 8 weeks of golf training in a centralized camp with identical accommodations and practice schedules.

The SMR group will perform supervised self-myofascial release exercises using Decathlon-brand foam rollers and balls, three times per week (30 min/session) in the gym after regular training.

The control group will engage in supervised 30-minute sessions of passive golf-related video watching, scheduled at the same time and environment as the SMR sessions.

Assessments will be conducted at Week 0 (baseline), Week 4 (midpoint), and Week 8 (post-intervention). Testing will include range-of-motion (ROM) measurements, balance tasks, strength/stability exercises, and golf swing performance using a TrackMan Launch Monitor. All outcome assessors will be blinded to group allocation to minimize bias.

The study aims to provide evidence on whether SMR is an effective training strategy to enhance functional movement and sports-specific performance in amateur golfers.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 18 to 25 years
* Collegiate golfers who are right-handed
* Currently active in university-level golf training (at least twice per week)
* Free of injuries or conditions that prevent participation in assessments or interventions
* Willing and able to provide written informed consent
* Not engaged in any other flexibility training or self-myofascial release (SMR) programs during the study period
* Exclusion Criteria:
* History of musculoskeletal injury or surgery within the past six months
* Diagnosed neurological disorders or balance impairments
* Current participation in other interventional studies
* Use of medications affecting neuromuscular function
* Any condition that prevents completion of golf swing or fitness testing

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Driver Club Head Speed | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Club head speed during driver shots was measured using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark) at a designated driving range. Participants were tested in groups of ten, using their own drivers (1-wood) for consistency. Prior to testing, each participant completed a supervised dynamic warm-up and five warm-up swings. They then performed five full-effort swings. Club head speed, defined as the velocity of the club head at ball impact, was recorded in miles per hour (mph). The average of the three most consistent shots (within 10% variance in ball flight) was used for analysis. All sessions were conducted at the same time of day under standardized environmental conditions, with new Titleist Pro V1 balls, fixed tee height, and pre-calibrated TrackMan settings.
Driver Carry Distance | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Carry distance for driver shots was measured using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark) at a designated driving range. All participants were tested in batches of ten and used their own 1-wood driver for consistency. Prior to testing, each participant completed a supervised dynamic warm-up and five warm-up swings. They then performed five full-effort swings. Carry distance was defined as the straight-line distance from the point of impact to where the ball first touched the ground, recorded in yards. The average of the three most consistent shots (with less than 10% variance in flight distance) was used for analysis. All tests were conducted under consistent environmental conditions (time of day, lighting, temperature) using standardized tee height and new Titleist Pro V1 balls. The TrackMan was recalibrated before each session.
Driver Side Deviation | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Driver side deviation was used to evaluate the lateral accuracy of tee shots with the driver (1-wood). Measurements were collected using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark), a radar-based device validated for golf performance analysis. Each participant used their personal driver to maintain equipment familiarity. After completing a standardized dynamic warm-up and five practice swings, participants executed five full-effort swings. Side deviation was defined as the absolute horizontal distance (in yards) between the ball's landing point and the intended target line, regardless of whether the miss was left or right. The three most consistent shots-those within a 10% variance in carry distance-were selected, and their average side deviation was calculated for analysis. Testing was conducted on the same designated driving range under consistent environmental conditions, including time of day, lighting, and temperature. New Titleist Pro V1 balls.
Driver Shot Proximity to Target | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Proximity to target was measured to assess the directional and distance accuracy of driver shots using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark). Each participant used their own 1-wood (driver) and performed five full-effort swings after completing a supervised dynamic warm-up and five warm-up swings. The test target was a fixed point on the driving range aligned with the intended launch line. Proximity was defined as the straight-line distance (in yards) between the ball's final landing position and the designated target. Among the five attempts, the three shots with the most consistent carry distances (within 10% variance) were selected for analysis, and the average proximity value was calculated. All tests were conducted at the same driving range location under standardized conditions, including consistent time of day, lighting, temperature, and wind. TrackMan was recalibrated before each session, and a standardized tee height and new Titleist Pro V1 balls.
Iron Club Head Speed | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Iron club head speed was measured using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark) to evaluate swing velocity during mid-iron shots. Participants used their own 7-iron club to ensure familiarity and consistency. Testing took place at a standardized driving range, with participants divided into batches of ten. Prior to data collection, each participant performed a supervised dynamic warm-up followed by five warm-up swings using their 7-iron. During testing, participants completed five full-effort swings. Club head speed was defined as the velocity of the club head at the exact moment of ball impact, expressed in miles per hour (mph). The average club head speed was calculated from the three most consistent shots, defined as those within a 10% variance in carry distance. All sessions were conducted at the same location and time of day under stable environmental conditions. The TrackMan device was recalibrated before each use, and standardized tee height and new Titlei
Iron Club Carry Distance | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Iron carry distance was measured using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark), a radar-based system commonly employed in golf performance analysis. Each participant used their personal 7-iron club to ensure comfort and familiarity. Testing was conducted at a consistent outdoor driving range setting, with participants grouped in batches of ten. Before testing, a standardized dynamic warm-up was completed under supervision, followed by five warm-up swings using the 7-iron. During the test, each participant performed five full-effort swings. Carry distance was defined as the horizontal distance the ball traveled through the air from the point of impact to its first landing point, measured in yards. For analysis, the average carry distance of the three most consistent shots-those falling within 10% variance in ball flight-was calculated. Testing was carried out at the same time of day under stable weather and lighting conditions to reduce variability.
Iron Club Side Deviation | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Iron side deviation was assessed using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark) to determine the lateral accuracy of 7-iron shots. Each participant used their own 7-iron club and performed five full-effort swings following a supervised dynamic warm-up and five preparatory swings. Side deviation was defined as the lateral distance in yards between the ball's landing point and the target line, irrespective of whether the deviation was left or right. For consistency, the three most accurate shots-defined as those with carry distance variation within 10%-were selected, and the average side deviation among them was calculated. Testing was conducted at the same outdoor driving range, in controlled environmental conditions (time of day, lighting, and temperature), and under supervision. Standardized tee height and new Titleist Pro V1 balls were used across all participants. The TrackMan device was recalibrated prior to each testing session to ensure measurement accuracy.
Iron Club Shot Proximity to Target | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Proximity for iron shots was measured using the TrackMan 3 Launch Monitor (TrackMan A/S, Vedbæk, Denmark) to assess target accuracy during 7-iron play. Each participant used their own 7-iron and performed five full-effort swings toward a designated pin positioned 130 yards away. Following a standardized dynamic warm-up and five warm-up swings, participants proceeded with the test. Proximity was defined as the straight-line distance from the ball's landing point to the center of the intended target. The three most accurate shots-based on consistent ball flight and carry distance within 10% variance-were selected, and their average proximity was calculated in yards. All tests were conducted at the same outdoor driving range under consistent environmental conditions (lighting, temperature, time of day), using new Titleist Pro V1 balls and fixed tee height. Testing was supervised by trained staff, and the TrackMan system was recalibrated before each session to ensure data precision.

SECONDARY OUTCOMES:
Ankle Dorsiflexion Range of Motion (Weight-Bearing Lunge Test) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Ankle dorsiflexion was assessed using the Weight-Bearing Lunge Test (WBLT), a reliable functional measure of closed-chain ankle range of motion. Participants stood facing a wall in a lunge position, with the test foot forward and heel flat on the ground. They were instructed to bend the front knee forward until it just touched the wall without lifting the heel. The distance from the longest toe to the wall was measured using a tape measure and recorded in centimeters. If maximal dorsiflexion was reached before the knee touched the wall, the angle between the tibia and vertical was measured using a digital inclinometer placed on the anterior tibia.Each participant completed two trials per leg, with the best score used for analysis. The test was administered barefoot under supervision to ensure consistent foot alignment and prevent compensatory movement.
Hip Flexion Range of Motion (Active, 90° Knee Flexion) | Week 0 (Pre-test): 1 day before the intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after the final SMR session
  Active hip flexion ROM was assessed with participants lying supine on a flat surface, maintaining the contralateral leg fully extended. Participants were instructed to actively lift the tested leg toward their chest, keeping the knee flexed at 90° throughout the motion. The measurement was taken at the point of maximum voluntary flexion, just before any compensatory pelvic movement was observed. A digital goniometer (e.g., Baseline® Digital Goniometer, accuracy ±1°) was positioned with the axis at the greater trochanter, the stationary arm aligned with the midline of the trunk, and the movable arm aligned with the lateral midline of the femur pointing toward the lateral epicondyle. Two trials were conducted, and the average value was used for analysis. All measurements were performed by the same trained tester to ensure reliability.
Hip External Rotation Range of Motion (Active, Seated, 90° Hip and Knee Flexion) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Active external rotation of the dominant hip was assessed in a seated position with both the hip and knee flexed at 90°, and the feet suspended off the ground. Participants were instructed to actively rotate the foot inward, thereby rotating the femur outward, as far as possible without leaning the trunk, lifting the thigh, or shifting weight. A digital goniometer (Lafayette Instrument Co., Model 01135, accuracy ±1°) was used for measurement. The axis was aligned with the center of the patella, the stationary arm was held perpendicular to the floor, and the movable arm followed the anterior midline of the lower leg, aligned with the tibial crest. Verbal instructions and light manual stabilization at the pelvis were used to prevent compensatory movement. Two trials were performed, and the average was recorded. All tests were conducted by the same trained examiner under standardized procedures.
Thoracic Spine Rotation Range of Motion (Active, Seated, Pelvis Stabilized) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Active thoracic spine rotation was measured with participants seated on a backless bench, hips and knees at 90°, feet flat on the floor, and arms crossed over the chest. The pelvis was stabilized using a fixed belt or manual support to isolate thoracic motion and prevent compensatory hip rotation. Participants were instructed to rotate their torso actively to the left and right as far as possible without leaning or flexing the spine. A digital goniometer (e.g., Baseline® Digital Goniometer, accuracy ±1°) was used to measure the angle between the initial and final positions of the shoulders relative to a fixed vertical axis. The average of two trials per direction was recorded. Testing was administered by the same trained evaluator under standardized conditions.
Shoulder Flexion Range of Motion (Active) | Week 0 (Pre-test): 1 day before the intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after the final SMR session
  Active shoulder flexion range of motion was assessed with participants lying supine. With the elbow extended and palm in a neutral position, each participant was instructed to actively lift the dominant arm in the sagittal plane toward the head, without arching the back or allowing scapular movement. A digital goniometer (Lafayette Instrument Co., Model 01135, accuracy ±1°) was used for measurement. The stationary arm was aligned with the mid-axillary line of the torso, the movable arm followed the lateral humerus toward the lateral epicondyle, and the axis was placed over the lateral aspect of the greater tubercle. To prevent compensatory lumbar extension, the evaluator provided verbal cues and light manual contact on the lower ribs. Two trials were conducted, and the average was used for analysis. All tests were completed by the same trained evaluator using standardized protocols to ensure measurement consistency.
Shoulder External Rotation Range of Motion (Active, Supine, 90° Abduction) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Active shoulder external rotation ROM was assessed with participants in a supine position, shoulder abducted to 90° and elbow flexed to 90°, with the upper arm supported on the table edge. Participants were instructed to actively rotate their forearm backward (external rotation) as far as possible without lifting the scapula or arching the back. A digital goniometer (Lafayette Instrument Co., Model 01135, ±1° accuracy) was used. The axis was placed on the olecranon, the stationary arm was perpendicular to the floor, and the movable arm aligned with the ulna. The examiner applied light manual contact on the anterior shoulder to prevent compensation. Two trials were recorded, and the average was used for analysis. All tests were performed by the same evaluator under standardized conditions.
Wrist Extension Range of Motion (Active, Seated, Neutral Forearm) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Active wrist extension ROM was measured with participants seated and their forearm in a neutral position (thumb up), elbow flexed at 90°, and hand over the table edge. Participants were instructed to extend their wrist upward as far as possible without moving their elbow, shoulder, or fingers. A digital goniometer (Lafayette Instrument Co., Model 01135, ±1° accuracy) was used. The axis was placed over the triquetrum, the stationary arm aligned with the ulna, and the movable arm along the fifth metacarpal. Two trials were recorded, and the average was used. A single trained evaluator conducted all tests under standardized conditions.
Single-Leg Stance Test (Eyes Closed) - Balance Time Measurement | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after the final SMR session
  Balance was assessed using the single-leg stance test with eyes closed. Participants stood barefoot on their dominant leg, arms crossed over the chest, and eyes gently closed. The non-stance leg was flexed at the knee so that the foot did not touch the ground. They were instructed to maintain balance as long as possible without moving the supporting foot, uncrossing their arms, or opening their eyes. The timing started once both eyes were fully closed and stopped when any of the following occurred: (1) the raised foot touched the ground, (2) arms moved from the chest, (3) the stance foot shifted, or (4) the eyes opened. A maximum time limit of 60 seconds was set. A stopwatch was used for timing, and one trained observer recorded each trial. Each participant performed two trials, and the longer duration was used for analysis. The same evaluator administered all tests to ensure consistency across sessions.
Rotational Medicine Ball Throw Distance (3kg, Standing Side Throw) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Rotational power and upper-body explosive strength were assessed using the Rotational Medicine Ball Throw Test. Participants stood on a flat, non-slip indoor surface with feet shoulder-width apart, holding a 3kg medicine ball at chest level with both hands. Maintaining an athletic stance with slight knee flexion, they were instructed to rotate the torso away from the throwing side and then explosively rotate toward the target, releasing the ball with maximal force in a side-throw motion toward a wall or open field area. Participants were instructed to keep both feet planted throughout the movement (no stepping or jumping was allowed). The distance from the throwing line to the point where the ball first contacted the floor was measured in meters. Each participant performed three valid throws, and the longest distance was recorded. A trained evaluator ensured correct form and consistency, counting only those throws that met the standard. Participants completed one practice trial before
Cross-Body Reach Test (High Plank, 30-Second Repetition Count) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Core coordination and shoulder stability were assessed using the Cross-Body Reach Test. Participants held a high plank position on a flat, non-slip indoor surface, with hands directly under the shoulders, elbows extended, and feet hip-width apart. Maintaining a straight line from head to heels, they were instructed to alternately lift one hand and tap the opposite shoulder (e.g., right hand to left shoulder), then return it to the ground, continuing the movement for 30 seconds.
  Each successful tap was counted as one repetition. The total number of valid repetitions performed within the 30-second period was recorded. A trained evaluator ensured correct form and consistency, counting only those repetitions that met the standard. Participants completed one practice trial before testing. This test emphasized neuromuscular control, core stability, and dynamic upper-limb coordination.
One-Repetition Maximum (1RM) Bench Press Test | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Upper body maximal strength was assessed using the One-Repetition Maximum (1RM) Bench Press Test. Participants lay supine on a flat, non-slip indoor bench, with feet flat on the floor, hands gripping the barbell slightly wider than shoulder-width apart, and elbows extended at the starting position. Maintaining stable torso alignment and controlled movement, they were instructed to lower the barbell until it lightly touched the chest (sternum level), pause briefly, then press the barbell back to full elbow extension. The load was progressively increased until the participant could no longer complete a valid repetition with proper form. The highest weight successfully lifted for one complete repetition was recorded as the 1RM value. A trained evaluator ensured correct technique and consistency, counting only those repetitions that met the standard. Participants completed one practice trial before testing. This test emphasized maximal upper-body strength, neuromuscular control, and movem
One-Repetition Maximum (1RM) Back Squat Test | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Lower body maximal strength was assessed using the One-Repetition Maximum (1RM) Back Squat Test. Participants stood on a flat, non-slip indoor surface, with the barbell placed across the upper trapezius (high-bar position), feet shoulder-width apart, and hands gripping the bar evenly. Maintaining a straight torso alignment and neutral spine, they were instructed to lower the body by flexing the hips and knees until the thighs were parallel to the floor or deeper, then return to the starting position by fully extending the hips and knees. The load was progressively increased until the participant could no longer complete a valid repetition with proper form. The highest weight successfully lifted for one complete repetition was recorded as the 1RM value. A trained evaluator ensured correct technique and consistency, counting only those repetitions that met the standard. Participants completed one practice trial before testing. This test emphasized maximal lower-body strength, neuromuscu
Pull-up Test (Maximal Repetition Count) | Week 0 (Pre-test): 1 day before intervention Week 4 (Mid-test): Day 28 ± 2 Week 9 (Post-test): 2 days after final SMR session
  Upper body muscular endurance was assessed using the Pull-up Test. Participants performed pull-ups on a standard fixed bar with an overhand (pronated) grip, hands placed slightly wider than shoulder-width apart. Starting from a dead hang position with arms fully extended and feet off the ground, they were instructed to pull the body upward until the chin cleared the bar, then lower back to the starting position in a controlled manner. Participants continued performing repetitions at a consistent pace until voluntary fatigue or failure to maintain proper form. Kipping, swinging, or using momentum was not permitted. Each valid repetition was counted toward the total score. The total number of correctly performed pull-ups without rest was recorded. A trained evaluator ensured correct form and consistency, counting only those repetitions that met the standard. Participants completed one practice trial before testing. This test emphasized upper-body muscular endurance, particularly in the

CONTACTS AND LOCATIONS:
Overall Officials: Kim Geok Soh, Professor, Study Director — Faculty of Educational Studies; Qi Yang, PHD, Principal Investigator — Faculty of Educational Studies
Locations (1):
- Hainan Normal University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality concerns, limited resources for data anonymization and management, and the scope of the study not requiring data sharing for external validation.

REFERENCES:
- See also: Provides details about the TrackMan 4 radar system used in this study to assess golf swing metrics such as club head speed and carry distance. — https://www.trackman.com/golf/launch-monitors/trackman-4?utm_source=chatgpt.com
- See also: Scientific article providing evidence that foam rolling interventions can improve joint range of motion-relevant to the theoretical basis of this trial. — https://pubmed.ncbi.nlm.nih.gov/26160309/